CLINICAL TRIAL: NCT05843682
Title: Technological Innovation in the Virtual Assistance of Patients With Uncontrolled Arterial Hypertension - Hyper 2
Acronym: Hyper2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Luiz Aparecido Bortolotto, Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5483/22/06
Record Dates: First submitted 2022-12-01; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Essential Hypertension; Metabolic Cardiovascular Syndrome; Heart Disease Risk Factors
Keywords: Remote telemonitoring; Uncontrolled hypertension; Artificial intelligent
MeSH Terms: conditions — Essential Hypertension; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatr (Other): In the inclusion visit, it will be install the Avatr App in the mobile device of the patients. The patients will give an evaluation to perform by the medical and nursing staff, where clinical data (office blood pressure, weight, height, abdominal circumference) will be collected and will answer questionnaires on quality of life, anxiety, sleep quality, food intake and therapeutic adherence. They will receive an automatic blood pressure measurement device to make household blood pressure measurement according to nursing guidance. Also, the patients will collected blood samples to further analysis for biochemical profile and 24-hour urine collection sample for urinary sodium dosage.
  The patients will take four in person visits after the initial visit, with the final visit after 12 months.
  Interventions: Device: Using the Avatr App
- Control (No Intervention): The patients will perform the same initial evaluation and answer the same questionnaires as described above for the Intervention Group. In this evaluation they will receive guidance regarding the adoption of life habits by the multidisciplinary team. The Control Group will receive reinforcement of guidance only in face-to-face visits.
  The patients will take four in person visits after the initial visit, with the final visit after 12 months.

INTERVENTIONS:
Device: Using the Avatr App — The patients will use the mobile application called Avatr, which will monitor their health data, as well as provide individualized care and early intervention through alerts generated for the multidisciplinary team.
  Arms: Avatr

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the use of artificial intelligence in home monitoring in patients with uncontrolled arterial hypertension.

DETAILED DESCRIPTION:
Arterial hypertension (AH) is one of the most important cardiovascular risk factors, accounting for 13.5% of all deaths worldwide. Mobile health technologies have been applied as an important tool to improve patient engagement and blood pressure (BP) control, as an alternative approach to remote monitoring of hypertensive patients. Therefore, it is essential to help patients adopt healthy measures to assist in the daily control of BP.

As the barriers to therapeutic adherence are complex and varied, solutions to improve adherence at the population level should be multifactorial. Therefore, the use of an application elaborated by artificial intelligence adapted to individual needs and customs, can help in improving therapeutic adherence and provide better bp control in patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion criteria:

1. Primary arterial hypertension in drug treatment with at least 3 classes of antihypertensive drugs in optimized dose
2. Aged between 20 and 65 years
3. Blood pressure of the office ≥ 140 and/or 90 mmHg
4. Facilities to use mobile and apps

Exclusion criteria:

1. Stroke sequelae
2. Cognitive dysfunction

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | One year
  Using the Avatr application with daily medication reminders, the patient will remember to use them. This way, there will be better control of blood pressure at home.
  Initially, 24-hour Ambulatory Blood Pressure Monitoring (ABPM) will be performed using the Spacelabs® device for initial control and during the four-monthly consultations, the mean blood pressure will be evaluated from the determination of systolic (SBP) and diastolic (DBP ) ) measured by an automatic sphygmomanometer (Omron HBP 1100 ®), on the right upper limb, with the individual sitting down, after 10 minutes of rest.
Glycemic control | One year
  Diabetic patients will have a personalized dietary guidance and will measure their blood glucose daily with the glucometer, in order to control the baseline blood glucose value.
Change of out-of-hospital visits | One year
  Change of extra-hospital visits during the monitoring period

SECONDARY OUTCOMES:
Patient engagement in treatment | One year
  To assess patient engagement, a structured questionnaire will be applied to verify the usability of the AVATR, as well as to obtain knowledge about how patients felt when using the application and the impact of this monitoring on their health.
Improvement in lifestyle | One year
  When performing daily physical activity after specialized evaluation and exercise prescription, with resistance and/or cardiovascular exercises, in addition to adhering to an adequate diet according to dietary guidelines, we can infer a reduction in weight (kg) and abdominal circumference (measurements in centimeter).

CONTACTS AND LOCATIONS:
Overall Officials: Fábio B Jatene, MD, PHD, Study Director — Heart Institute
Locations (1):
- Heart Institute (InCor), Hospital das Clinicas do HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dupont J, Dupont JC, Milon H, Froment A. [Spontaneous mortality and vascular lesions in 3 rat strains with different blood pressure levels]. C R Acad Hebd Seances Acad Sci D. 1975 Apr 7;280(13):1637-40. French. PMID 152
- See also: PubMed Single Citation Matcher — https://pubmed.ncbi.nlm.nih.gov/?term=Bortolotto%2C+LA%5BAuthor%5D

DOCUMENTS (2):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT05843682/Prot_000.pdf
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT05843682/ICF_001.pdf